CLINICAL TRIAL: NCT03476954
Title: Perfusion Enhancement With Respiratory Impedance in Stroke (PERI-Stroke)
Acronym: PERI-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Steven Messe, Associate Professor of Neurology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 824558
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory impedance monitoring session (Experimental)
  Interventions: Other: Respiratory Impedance (RI)

INTERVENTIONS:
Other: Respiratory Impedance (RI) — A non-invasive respiratory device is employed to generate resistance during the inspiratory phase of respiration.

SUMMARY:
This is a non-randomized phase 2 study designed to asses the mean flow velocity (MFV) and cerebral blood flow (CBF) response to non-invasive respiratory impedance.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Ability and willingness to sign informed consent by patient or legally acceptable surrogate decision maker
3. Acute ischemic stroke within 72 hours of study enrollment
4. Imaging or examination confirming unilateral frontal lobe involvement in the stroke

Exclusion Criteria:

1. Hemorrhagic conversion of ischemic infarct
2. History or presence of congestive heart failure, as defined by any of the following:

   1. Any preceding diagnosis of congestive heart failure as per patient report or medical record
   2. Report of moderate or severe systolic or diastolic dysfunction on prior
   3. Reduced ejection fraction, <50%, on prior echocardiogram
   4. Jugular venous pulsations >10 cm
   5. Pulmonary edema on chest radiography Of note, an echocardiogram is not required prior to study enrollment.
3. History or presence of cardiomyopathy, as per medical record, patient report, or prior echocardiogram
4. History or presence of pneumothorax or hemothorax
5. History or presence of COPD
6. History of current use of home oxygen
7. Presence of pneumonia, as clinically determined by the primary medical team after admission chest radiography
8. Age < 18 years
9. Skull defect that would interfere with CBF monitoring
10. Pregnancy (urine or serum testing will required prior to enrollment of any pre-menopausal women)
11. Structural brain lesion, including known primary tumor, metastatic tumor, or vascular malformation
12. Prior neurosurgical procedure
13. Any medical condition that the clinical investigator feels would pose a hazard to the subject if he/she participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in CBF that occurs during RI, as measured by diffuse correlation spectroscopy (DCS) with a sampling frequency of 5 Hz | Baseline
Reports of any of the following: shortness of breath, chest pain, fatigue, or hypoxia | Baseline

SECONDARY OUTCOMES:
Change in MFV as measured by transcranial doppler (TCD), during RI | Baseline
Change in mean arterial pressure (MAP,) during RI | Baseline
Change in end-tidal carbon dioxide (CO2), during RI | Baseline
Time to maximum CBF effect after the introduction of RI | Baseline
Change in National Institute of Health Stroke Scale (NIHSS) (admission vs discharge) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No